CLINICAL TRIAL: NCT06831214
Title: Assessment of Bone Gain Following Composite Graft Rehabilitation of Horizontal Maxilla Atrophy With Sausage Technique Utilizing (Pericardial) Collagen Membrane Versus Periosteal Membrane Harvested From the Iliac Crest A Randomized Clinical Trial
Brief Title: Assessment of Bone Gain Following Composite Graft Rehabilitation of Horizontal Maxilla Atrophy With Sausage Technique Utilizing (Pericardial) Collagen Membrane
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Manaf Omar Alhabshi, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-25
Record Dates: First submitted 2025-01-30; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Maxilla Atrophy
Keywords: collagen membrane; Periosteal membrane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pericardial collagen membrane (Experimental): Sausage Technique: Specifically designed for cases with severely thin ridges, this technique utilizes a collagen membrane stabilized with titanium pins to secure the bone graft. This helps prevent the migration or collapse of graft particles, promoting better bone gain and healing
  Interventions: Other: (pericardial) collagen membrane
- periosteal Membrane harvested from anterior iliac bone (Active Comparator): The choice of comparators in clinical studies involving guided bone regeneration (GBR) often includes both nonresorbable and resorbable membranes. Resorbable membranes have demonstrated better soft tissue compatibility compared to nonresorbable options, making them a preferred choice in many cases. For instance, studies have shown that using an organic bovine bone-derived mineral (ABBM) in conjunction with a rapidly resorbing natural collagen membrane is effective for horizontal ridge augmentation, as evidenced by positive histologic outcomes.
  Interventions: Other: periosteal Membrane harvested from anterior iliac bone

INTERVENTIONS:
Other: (pericardial) collagen membrane — bone gain following composite graft rehabilitation of horizontal maxilla atrophy with sausage technique utilizing (pericardial) collagen membrane
  Arms: pericardial collagen membrane
Other: periosteal Membrane harvested from anterior iliac bone — The choice of comparators in clinical studies involving guided bone regeneration (GBR) often includes both nonresorbable and resorbable membranes. Resorbable membranes have demonstrated better soft tissue compatibility compared to nonresorbable options, making them a preferred choice in many cases. For instance, studies have shown that using an organic bovine bone-derived mineral (ABBM) in conjunction with a rapidly resorbing natural collagen membrane is effective for horizontal ridge augmentation, as evidenced by positive histologic outcomes.
  Arms: periosteal Membrane harvested from anterior iliac bone

SUMMARY:
This study designed to assess amount of bone gain following composite graft rehabilitation of horizontal maxilla atrophy with sausage technique utilizing (pericardial) collagen membrane versus Periosteal membrane harvested from the iliac crest in 6 months.

DETAILED DESCRIPTION:
Edentulous Maxillary ridges are a growing challenge worldwide. According to a fact sheet released by the World Health Organization (WHO) in 2022. teeth loss can be attributed to many conditions, mainly advanced dental caries, and severe periodontal disease. But pathology trauma and infection are other potential causes. Substantial studies have shown Dental implants as an excellent treatment choice with predictable long-term results.

However, to guarantee the success of implant stability at the time of insertion, a sufficient amount of bone width is robust. As known that bone surrounding extracted teeth resorb in all directions. This leads to horizontal and vertical bone volume loss reaching up to 50% in width reduction which compromises dental implant insertion. Cawood and Howell in 1988 categorized the degrees of edentulous ridge atrophy into six categories, emphasizing category IV atrophies which are known as "knife-edge" ridge, present a serious horizontal defect, making dental implant placement a challenge.

The challenge of bone defects augmentation primarily lies in the insufficient bone volume at the implant site, which can negatively impact the success of dental implants. Severe horizontal bone defects, such as those classified as "knife-edge" ridges, present significant obstacles for effective implant placement. Sausage Technique: Specifically designed for cases with severely thin ridges, this technique utilizes a collagen membrane stabilized with titanium pins to secure the bone graft. This helps prevent the migration or collapse of graft particles, promoting better bone gain and healing. Still some limitation of this technique including possibility of the collagen membrane becoming exposed during the healing process, which can compromise the regenerative outcome. Limited Bone Gain: In some cases, the amount of bone gain achieved may not meet the expectations, particularly in severely atrophic ridges, which can lead to the need for additional augmentation procedures. A study by Fernando V, et al showed that recipient sites augmented with autogenous bone grafts and preserved periosteal membranes maintained an average bucco-lingual width of 8.1 mm after augmentation, which was significantly greater than the baseline width of 3.2 mm. This augmented width was maintained at 98% after an average follow-up of 2.9 years. Another study by Kubota and Shirasuna evaluates the effectiveness of free periosteum in secondary bone grafting for maxillary alveolar clefts.

Results indicate that 97.1% of patients receiving free periosteum achieved significant vertical bone formation, compared to 79.5% in the control group. While the free-periosteum group experienced a higher rate of postoperative wound dehiscence. The rationale of the study is to evaluate the effectiveness of a combination of autogenous bone and an organic bovine bone-derived mineral (ABBM) for horizontal ridge augmentation using sausage technique utilizing (pericardial) collagen membrane versus Periosteal membrane harvested from the iliac crest. The study aimed to Assess bone gain in insufficient maxillary alveolar ridge width, particularly in patients with knife-edge ridges, to facilitate successful dental implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Age range (18-60 years)
* Patients with unilateral or bilateral horizontal atrophy in maxilla with minimum 1 quadrant.
* No intervention done previously on the donor and host sides.
* No sex predilection

Exclusion Criteria:

* Syndromic patients.
* bone metabolism & systemic diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Horizontal bone gain | 6 months
  Bone caliper intra-operative and at time of implant placement CBCT, preoperative, immediate to assess amount of bone gain postoperative

SECONDARY OUTCOMES:
Percentage of newly formed bone | 6 months
  Bone core biopsy from the augmentation site with Histomorphometric analysis to assess amount of bone gain

CONTACTS AND LOCATIONS:
Overall Officials: Manaf O Alhabshi, Msc, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No